CLINICAL TRIAL: NCT00502359
Title: Testing Ascensia Contour Glucometer for the Measurement of Blood Glucose Values in Pregnancy
Brief Title: Testing Ascensia Contour Glucometer for the Measurement of Blood Glucose
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Bayer (Industry)
Other Study IDs: keinen
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes, screening, glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: capillary blood glucose measurement

SUMMARY:
Present practice: Measurement of fasting glucose values in 2nd trimester of pregnancy, if above 4.8 mmol/l, a Glucose Tolerance Test is performed. (Two-step procedure: 1. Appointment for the fasting glucose measurement, 2. Appointment for the Glucose Tolerance Test)

DETAILED DESCRIPTION:
Present practice: Measurement of fasting glucose values in 2nd trimester of pregnancy, if above 4.8 mmol/l, a Glucose Tolerance Test is performed. (Two-step procedure: 1. Appointment for the fasting glucose measurement, 2. Appointment for the Glucose Tolerance Test) Study: Testing of reliability and applicability of the Ascensia Contour Glucometer, Bayer. Comparison of 100 fasting glucose values measured in venous plasma by the hexokinase method in the Laboratory with 100 fasting glucose values measured in capillary whole blood on the Ascensia Contour Glucometer Outcome: If Ascensia Contour Glucometer shows applicable accuracy (narrow scatter of values), the two-step procedure should be replaced by one-step procedure: 1 only one appointment for the measurement of the fasting glucose value in capillary whole blood on Ascensia Contour Glucometer and if above 4.8 mmol/l Glucose Tolerance Test on the same day

ELIGIBILITY:
Inclusion criteria:

* Healthy pregnant women in 2nd Trimester of pregnancy scheduled for the measurement of fasting glucose value

Exclusion criteria:

* Pregnant women with pre-existent (Type 1 or 2) diabetes or already diagnosed diabetes of pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2005 (Actual)
Dates: Start 2005-04; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Clinic of obstetrics, University Hospital of Zurich, Zurich, Switzerland